CLINICAL TRIAL: NCT04289025
Title: Digital Health: Modelling and Artificial Intelligence Using Sensor Data to Personalise REHABilitation Following Joint Replacement
Brief Title: Modelling and AI Using Sensor Data to Personalise REHABilitation Following Joint Replacement
Acronym: MAPREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: Dynamic Metrics Ltd (Industry); University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dig Health01
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Arthroplasty Complications
Keywords: Arthroplasty; Replacement Rehabilitation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Personalised exercise programme is provided to the exercise group.
  Interventions: Other: Exercise
- No Intervention (No Intervention): This group of patients will receive no intervention.

INTERVENTIONS:
Other: Exercise — A set of exercises are provided to each patient.
  Arms: Exercise

SUMMARY:
This study aims to determine a volunteer's gait objectively after surgery, when signed off from the consultant and physiotherapist. This will identify any gait deficiencies using simple traffic light coding, using GaitSmart, a CE Marked Class 1M Medical Device. Volunteers chosen for the intervention programme, a set of exercises to improve gait deficiencies identified in the report. All the exercises will be standard one already used within the NHS. The objectives are to compare the outcomes from the intervention group with the Standard of Care group, in terms of gait and PROMS and from this determine the clinical and economic benefits of the intervention.

DETAILED DESCRIPTION:
This study aims to determine a volunteer's gait objectively after surgery, when signed off from the consultant and physiotherapist. This will identify any gait deficiencies using simple traffic light coding, using GaitSmart, a CE Marked Class 1M Medical Device. All volunteers in the intervention group will be provided with a copy of their report. Protocol for SoC group SoC volunteers receive a GaitSmart test at their first appointment but are not given their report. Questionnaires to record Volunteer reported outcome measures (PROMS) include: Oxford hip score (OHS) or Oxford knee score (OKS) plus the Euroqol questionnaire (EQ5D-5D) are completed. SoC volunteers return at week 15 for a second test but are not given their report. Questionnaires to record Volunteer reported outcome measures (PROMS) include: Oxford hip score (OHS) or Oxford knee score (OKS) plus the Euroqol questionnaire (EQ5D-5D) are completed. Protocol for GaitSmart intervention group GaitSmart intervention group have the procedure explained to them at the first appointment. All exercises have the volunteer standing or sitting and are chosen from exercises already provided by the NHS. Each volunteer will get a subset of these. The nurse will ensure volunteers can perform the exercises before leaving the session. GaitSmart test performed at weeks 6, 9, 12 and 15. The report is provided plus six personalised exercises. The nurse will check they are able to perform the tests at each visit. Those not suitable will be struck off the list. Questionnaires to record Volunteer reported outcome measures (PROMS) will be completed at weeks 6 and 15.

ELIGIBILITY:
Inclusion:

1. The subject must provide written informed consent.
2. Subject is scheduled for primary Total Knee replacement / Total Hip replacement within the next 30 days.
3. Subject is considered skeletally mature.
4. Subject is willing, able, and plans to perform the activities associated with the study.
5. Unilateral or bilateral hip or knee replacement volunteers free of moderate to severe pain in the contralateral limb.
6. Signed off at 6 weeks by physiotherapist.

Exclusion:

1. Will not be a resident living within the catchment area for Norfolk & Norwich University hospital for at least 6 months post-surgery.
2. Undertaking the surgery as a private patient.
3. Patients who, in the opinion of the clinical staff, do not have capacity to consent.
4. Patients who are pregnant.
5. Unable to understand written and spoken English.
6. Patient who is currently enrolled in another interventional trial involving surgery, exercise or rehabilitation.
7. Any neurological condition that affects movement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Objective change in gait kinematics | 15 weeks post op
  Change in a patient's gait measured objectively using Gaitsmart
Subjective change in gait | 15 weeks post op
  Change in a patient's Oxford hip or knee score
Quality of life changes | 15 weeks post op
  Change in a patient's Quality of Life score (EQ5D)

CONTACTS AND LOCATIONS:
Overall Officials: Iain McNamara, MD, Principal Investigator — Clinical Research and Trials Unit (Norfolk and Norwich University Hospital, UK)
Locations (1):
- Norfolk and Norwich University Hospital, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared by all partners. Only Norfolk and Norwich University Hospital will hold full patient data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 0 to 28 months, which is 12 months after project completion.
Access Criteria: Access to the research dataset will be permitted via application to the CI's and sponsor.